CLINICAL TRIAL: NCT05603013
Title: Vinorelbine Metronomic Chemotherapy Combined With Hypofractionated Radiotherapy, PD-1/PD-L1 Inhibitor Sequential GM-CSF and IL-2 for Treatment of Advanced Refractory Non-small Cell Lung Cancer and Breast Cancer (PRaG 6.0)
Brief Title: Vinorelbine Metronomic Chemotherapy Combined With Hypofractionated Radiotherapy, PD-1/PD-L1 Sequential GM-CSF and IL-2 for Treatment of Advanced Refractory Non-small Cell Lung Cancer and Breast Cancer(PRaG 6.0)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2022-136-01
Record Dates: First submitted 2022-10-29; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma Breast
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Vinorelbine; Radiotherapy; Immune Checkpoint Inhibitors; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vinorelbine Combined With Radiotherapy, PD-1/PD-L1 Sequential GM-CSF and IL-2 (Experimental): Vinorelbine Metronomic Chemotherapy Combined With Hypofractionated Radiotherapy, PD-1/PD-L1 Sequential GM-CSF and IL-2
  Interventions: Drug: Vinorelbine; Radiation: Radiotherapy; Drug: PD-1/PD-L1 inhibitor; Drug: GM-CSF; Drug: IL-2

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine Tartrate Oral
Radiation: Radiotherapy — hypofractionated radiotherapy
Drug: PD-1/PD-L1 inhibitor — PD-1/PD-L1 inhibitor subcutaneous injection or intravenous injection
Drug: GM-CSF — GM-CSF subcutaneous injection
Drug: IL-2 — IL-2 subcutaneous injection

SUMMARY:
This is an open-label, single-arm, Phase II investigator-initiated trial of vinorelbine metronomic chemotherapy combined with hypofractionated radiotherapy, PD-1/PD-L1 inhibitor sequential GM-CSF and IL-2 for treatment of advanced refractory non-small cell lung cancer and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and above;
2. Diagnosed with histologically or cytologically-confirmed, standard treatment is ineffective (disease progresses after treatment) or locally advanced or metastatic malignant non-small cell lung cancer and breast cancer patients who cannot tolerate standard therapy, cannot receive or do not have standard therapy;
3. ECOG(Eastern Cooperative Oncology Group) performance is 0-3;
4. Life expectancy greater than 3 months;
5. T lymphocyte absolute value ≥0.5 upper limit of normal (ULN), absolute neutrophil count(ANC)≥1.0 x 10(9)/L#serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3.0*ULN, or AST and ALT≤5*ULN with hepatic metastasis; Total serum creatinine ≤1.5*ULN#
6. Signed informed consent form# -

Exclusion Criteria:

1. Current pregnancy or lactation# 2. History of other malignant tumors within 5 years prior to dose administration, expect for#malignancies that can be cured after treatment (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer); 3. Uncontrolled epilepsy, central nervous system diseases or mental illness; 4. Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or greater than or equal to Class 2 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study; 5. Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation; 6. Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interpretation of outcomes, including active opportunistic infections or advanced (severe) infections, uncontrolled diabetes; 7. Allergic to any of the ingredients used in the study; 8. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation, or other immune-related disease requiring long-term oral hormone therapy; 9. Acute and chronic tuberculosis infection; 10. Other disorders with clinical significance according to the researcher's judgment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate #ORR# | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 24 months
  PFS was defined as the time from the first administration of study treatment to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever comes first.
Disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants with a complete response (CR), partial response (PR), or stable disease (SD)
Overall survival (OS) | 24 months
  OS was defined as the time from the first administration of study treatment to death from any cause.
Adverse event | 24 months
  rate of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No